CLINICAL TRIAL: NCT00000809
Title: A Phase I Trial of the Safety and Immunogenicity of MN rsgp120/HIV-1 With the Adjuvants QS-21 and Alum Compared to MN rsgp120/HIV-1 and QS-21 in Infants Born to HIV-Infected Women
Brief Title: Safety and Effectiveness of Two Different Formulations of an HIV Vaccine in Infants Born to HIV-Infected Women
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Prevention
Other Study IDs: ACTG 279; 11255 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; HIV Seronegativity
Keywords: HIV Preventive Vaccine; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections | interventions — Aluminum Hydroxide; saponin QA-21V1

INTERVENTIONS:
Biological: Aluminum hydroxide
Biological: QS-21
Biological: MN rsgp120/HIV-1

SUMMARY:
The purpose of this study is to test the safety and effectiveness of two different formulations of an HIV vaccine in infants born to HIV-infected women.

ELIGIBILITY:
Inclusion Criteria

Infants may be eligible for this study if they:

* Are 1 to 3 days old.

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)